CLINICAL TRIAL: NCT01699620
Title: Evaluation of Soft Tissue Healing and Implant Stability of Cochlear Baha BI300 Implants Loaded From 2 Weeks Post-surgery: a Comparison Between Two Surgical Techniques.
Brief Title: Comparative Study of Two Surgical Techniques for Soft Tissue Healing and Implant Stability of Cochlear BI300 Implants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Denmark: Danaflex A/S, national distributor of Cochlear Ltd (Unknown)
Responsible Party: Principal Investigator, Dr. Lars Vendelbo Johansen, MD, DMSc, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66.20.19.1.LV
Record Dates: First submitted 2012-09-25; First posted 2012-10-03 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Hearing Loss, Conductive
Keywords: Bone anchored hearing aid; Soft tissue healing; Implant stability; Linear incision; Dermatome technique; Hearing Aids; Implants, Artificial; Surgical Procedures, Operative
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermatome (Experimental): BAHA implant insertion with Dermatome technique
  Interventions: Procedure: BAHA implant insertion
- Linear incision (Experimental): BAHA implant insertion with linear incision
  Interventions: Procedure: BAHA implant insertion

INTERVENTIONS:
Procedure: BAHA implant insertion — The intervention is insertion of the Cochlear Bi300 to be used for bone anchored hearing aid.
  Other Names: Cochlear Bi300

SUMMARY:
The study compares two different operative techniques for placement of the Cochlear Bi300 implant to be used for bone anchored hearing aid. The operative techniques to be compared are

* Dermatome technique with soft tissue reduction
* Linear incision with minimal or no soft tissue reduction

The hypothesis is that the operative techniques are comparable with regard to implant stability, soft tissue healing and loss of sensibility around the implant.

To evaluate the evolution of implant stability during the early healing period after implantation, which is the most critical period for osseointegrated implants, in particular when early loading protocols are used.

To compare soft tissue healing around Baha implants placed according to the recommended surgical technique with skin transplant and Baha implants without performing skin reduction.

To compare the loss of sensibility of the skin around the Baha implant (some loss of cutaneous sensibility nerves in the transplant procedure) between the two surgical procedures.

While the study focuses on the early healing period (3 months), long-term safety data will also be collected after 6 months and 1-year.

The study will also evaluate the change in health status produced by the surgical intervention.

DETAILED DESCRIPTION:
1. BACKGROUND

   Implant stability

   Until recently, the implants used in Baha surgery have exclusively been standard Brånemark type of titanium implants with an as-machined surface finish. The recommended procedure for Baha implantation with the machined titanium implants uses a 12-week healing period before loading the implant with a sound processor, in order to allow sufficient time for the implant to become integrated in the bone. The new Cochlear Baha BI300 Series implant has been designed to improve implant stability at placement and over time, thus making it possible to reduce the time to sound processor fitting. The implant features a wider diameter compared to the previous generation Baha implant, small-sized threads at the cylindrical portion of the implant underneath the flange, and a roughened implant surface.

   Six-month data from a multi-centre clinical investigation comparing the new implant with the previous generation Baha implant using a 6-week loading protocol, shows significantly higher Implant Stability Quotient (ISQ) values (measured by resonance frequency analysis) for the new implant at each time point, and no reduction in stability after loading.1 The data from the study suggest that the implant stability achieved 6 weeks after implantation is sufficient to support the sound processor. The data also suggest that a further reduction of the time to sound processor fitting may be possible, provided favourable bone conditions at the implant site and provided satisfactory soft tissue status at the time of loading. Hence, a clinical investigation with implant loading 21 days post-surgery was initiated by the team in Nijmegen, and 6-month data from the investigation confirm that it is safe to attach the sound processor after 3 weeks.2 Early results from two other studies using loading times of 4 weeks3 and 2 weeks4, respectively, have also been presented and show good outcomes. All studies have been performed on patients with good bone quality.

   Soft tissue management

   The recommended procedure for Baha implantation advocates a hair free transplant measuring 25 x 25 mm placed direct on the periosteum. The purpose is to obtain an immobile skin, hence reducing the risk of adverse skin reactions in the area. Since there is no or only weak adherence between the titanium abutment and surrounding soft tissue it is anticipated that, if no skin reduction is performed, epidermal downgrowth and pocket formation may occur over time, increasing the risk for infection in the implant area. The current surgical procedure, with skin transplant, has been used for three decades and proven safe; however, skin complications still occur and account for the majority of reported complications with Baha implants.

   Some surgeons have hypothesised that equally good or better results may be achieved if the soft tissue is left intact. However, the clinical evidence still remains scarce and a systematic follow-up is lacking. To the investigators knowledge, the only publication specifically focusing on the alternative surgical technique without soft tissue thinning is a limited study by Dr. Hultcrantz comparing outcomes in seven patients undergoing Baha surgery with the traditional surgical technique (with skin thinning) and seven patients with the alternative technique (without skin thinning).5 The outcomes of the study are promising, but more clinical data is necessary to establish whether the surgical technique is safe and efficacious.
2. OBJECTIVES

To evaluate the evolution of implant stability during the early healing period after implantation, which is the most critical period for osseointegrated implants, in particular when early loading protocols are used.

To compare soft tissue healing around Baha implants placed according to the recommended surgical technique with skin transplant and Baha implants without performing skin reduction.

To compare the loss of sensibility of the skin around the Baha implant (some loss of cutaneous sensibility nerves in the transplant procedure) between the two surgical procedures.

While the study focuses on the early healing period (3 months), long-term safety data will also be collected after 6 months and 1-year.

The study will also evaluate the change in health status produced by the surgical intervention.

6. IMPLANT DEVICE

The following CE marked implant with pre-mounted abutment shall be used (MDD Class IIb medical devices, manufacturer: Cochlear Bone Anchored Solutions AB, Mölnlycke, Sweden):

• Cochlear Baha BIA300 Implant 4 mm with Abutment 9 mm (Article # 92346)

Note: The 9 mm abutment will be used in both treatment groups (with and without skin transplant) in order to be able to compare results from resonance frequency analyses (implant stability) during the early healing period. When appropriate, the patients with skin reduction will have the 9 mm abutment exchanged to a 6 mm abutments (Article # 92130) after 3-month data has been collected. No further surgery is needed in order to exchange the 9 mm abutment to 6 mm abutment.

7. TREATMENT

Implantation and use of the Baha system (hearing device/implant system). The implants shall be placed according to the procedure for FAST (one-stage) surgery.

All patients will receive treatment, thus no placebo control group is used.

8. METHOD

This evaluation will be performed at one site. Implants will be placed in a one-stage surgical procedure. Sound processor fitting will be performed 2 weeks after implant installation, or at the discretion of the investigator. The decision to load an implant will be based on assessment of implant stability and status of the soft tissue. Patients who are evaluated as not ready to be loaded 2 weeks after surgery will be loaded as soon as the healing is sufficient.

Patients included in the study will be randomised into two different treatment groups where the patients in one group will have soft tissue removed and split skin (harvested with dermatome) will be used to cover the periosteum around the abutment as per the recommended procedure by the manufacturer, and the patients in the other group will not have any soft tissue removed (a linear incision technique will be used). If the subcutaneous tissue is of a thickness so that it is not possible to use a 9 mm abutment, minimal removal of the subcutaneous tissue superficial of the fascia will be performed.

The risks with this treatment are the same for the two treatment groups and are: bleeding per- and postoperatively, wound infection and damage to surrounding tissues including sensory nerves to the scalp and loss of the implant. These risks are well known risks with known treatments. The new surgical procedure does not introduce any new risks.

The change in health status produced by the surgical intervention is evaluated with the Glasgow Benefit Inventory 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss suitable for bone anchored hearing aid
* Capable of maintaining sufficient hygiene around the implant.

Exclusion Criteria:

* Previous radiotherapy to the operation area
* Diabetes
* Skin disease in the operation area
* Any relevant medical history or current disease/treatment/medication that may affect bone or skin quality in the implant area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Implant stability, day of surgery | Day of surgery
  Implant stability shall be assessed using resonance frequency analysis. The measurement renders Implant Stability Quotient (ISQ) values from 1 to 100. Two perpendicular measurements shall be performed at each implant. The highest and lowest ISQ value out of three measurements obtained at each time point shall be recorded. Measurements shall be performed at the abutment level, and the Osstell ISQ instrument and SmartPeg Type 55 (Osstell, Gothenburg, Sweden) shall be used.
  Note: If a patient requires a change of abutment height, ISQ values shall be recorded on both abutment heights at the time of abutment change, in order to obtain a reference value for subsequent RFA measurements.
Implant stability, early healing phase | 3 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, early healing phase | 7 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, early healing phase | 10 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, loading of implant | 14 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, middle healing phase | 21 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, middle healing phase | 30 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, late healing phase | 60 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, late healing phase | 180 days postoperatively
  See description for "Implant stability, day of surgery".
Implant stability, late healing phase | 1 year postoperatively
  See description for "Implant stability, day of surgery".

SECONDARY OUTCOMES:
Soft tissue status | 3 days postoperatively
  The status of the soft tissue around the abutment shall be assessed using the classification proposed by Holgers et al, referred to as Holgers Index. See scale below:
  Grade 0 No irritation. Epidermal debris removed if present. Grade 1 Slight redness. Temporary local treatment. Grade 2 Red and slightly moist tissue. No granulation formation. Local treatment, extra controls.
  Grade 3 Reddish and moist. Sometimes granulation tissue. Revision surgery is indicated.
  Grade 4 Removal of skin-penetrating implant or abutment necessary due to infection.
  Grade R Removal of implant for reasons not related to skin problems.
Soft tissue status | 7 days postoperatively
  See "Soft tissue status" - 3 days postoperatively
Soft tissue status | 10 days postoperatively
  See "Soft tissue status" - 3 days postoperatively.
Soft tissue status | 14 days postoperatively
  See "Soft tissue status" - 3 days postoperatively.
Soft tissue status | 21 days postoperatively
  See "Soft tissue status" - 3 days postoperatively.
Soft tissue status | 30 days postoperatively
  See "Soft tissue status" - 3 days postoperatively.
Soft tissue status | 60 days postoperatively
  See "Soft tissue status" - 3 days postoperatively.
Soft tissue status | 180 days postoperatively
  See "Soft tissue status" - 3 days postoperatively.
Soft tissue status | 1 year postoperatively
  See "Soft tissue status" - 3 days postoperatively.

OTHER OUTCOMES:
Loss of implant | 12 months
  Every loss of implant will be recorded and reported to the manufacturer.
Change in health status | 3 months
  The change in health status produced by the surgical intervention is evaluated with the Glasgow Benefit Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Vendelbo Johansen, MD, DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, ENT-department, Aarhus, Denmark

REFERENCES:
- [Background] Dun CA, de Wolf MJ, Hol MK, Wigren S, Eeg-Olofsson M, Green K, Karlsmo A, Flynn MC, Stalfors J, Rothera M, Mylanus EA, Cremers CW. Stability, survival, and tolerability of a novel baha implant system: six-month data from a multicenter clinical investigation. Otol Neurotol. 2011 Aug;32(6):1001-7. doi: 10.1097/MAO.0b013e3182267e9c. PMID 21725257
- [Background] Dun CAJ, Faber HT, Mylanus EA, Cremers CW, Hol MK. Implant stability after earlier loading of the Baha BI300 implant. Proceedings of the Third International Symposium for Bone Conduction Hearing - Craniofacial Osseointegration; 2011 Mar 23-26; Sarasota, USA.
- [Background] McLarnon C, Johnson I, Davison T, Hill J, Henderson B, Leese D, Morley D. Evidence for early loading of Baha BI300 system at four weeks. Proceedings of the Third International Symposium for Bone Conduction Hearing - Craniofacial Osseointegration; 2011 Mar 23-26; Sarasota, USA.
- [Background] Green KM, Exley RP, Bruce IA, Andrew R. First experiences of loading a Baha sound processor at 2 weeks following surgery. Presented at the Third International Symposium for Bone Conduction Hearing - Craniofacial Osseointegration in Sarasota, USA, 23-26 March 2011
- [Background] Hultcrantz M. Outcome of the bone-anchored hearing aid procedure without skin thinning: a prospective clinical trial. Otol Neurotol. 2011 Sep;32(7):1134-9. doi: 10.1097/MAO.0b013e31822a1c47. PMID 21817939
- [Background] Holgers KM, Tjellstrom A, Bjursten LM, Erlandsson BE. Soft tissue reactions around percutaneous implants: a clinical study of soft tissue conditions around skin-penetrating titanium implants for bone-anchored hearing aids. Am J Otol. 1988 Jan;9(1):56-9. PMID 3364537
- [Background] Robinson K, Gatehouse S, Browning GG. Measuring patient benefit from otorhinolaryngological surgery and therapy. Ann Otol Rhinol Laryngol. 1996 Jun;105(6):415-22. doi: 10.1177/000348949610500601. PMID 8638891